CLINICAL TRIAL: NCT00894400
Title: Characterisation of Fractionated Electrograms Critical for Maintenance of AF
Brief Title: Characterisation of Fractionated Electrograms Critical for Maintenance of Atrial Fibrillation (AF)
Acronym: CAFE AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Dr Richard Schilling, Barts and The London NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0703/6
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: Atrial Fibrillation
Keywords: AF; catheter ablation; fractionated electrogram; complex fractionated atrial electrogram (CFAE)
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeting of most fractionated electrograms first (Experimental): During catheter ablation of AF patients will have fractionated electrograms targeted. In the experimental group the fractionated electrograms believed to be most critical will be targeted first.
  Interventions: Procedure: catheter ablation
- Targeting least fractionated electrograms first (Active Comparator): During catheter ablation of AF fractionated electrograms are targeted. In this arm the least fractionated electrograms will be targeted first.
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: catheter ablation — catheter ablation using radiofrequency energy

SUMMARY:
The purpose of this study is to characterise which fractionated electrogram morphologies are important to target in the catheter ablation of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* patients with persistent AF listed for first time catheter ablation

Exclusion Criteria:

* age < 18 years
* pregnancy
* contraindications to procedure
* recent myocardial infarction, coronary intervention, or cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
change in AF cycle length when targeting fractionated electrograms of different morphology. | immediate

CONTACTS AND LOCATIONS:
Locations (1):
- Barts and The London NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Hunter RJ, Diab I, Tayebjee M, Richmond L, Sporton S, Earley MJ, Schilling RJ. Characterization of fractionated atrial electrograms critical for maintenance of atrial fibrillation: a randomized, controlled trial of ablation strategies (the CFAE AF trial). Circ Arrhythm Electrophysiol. 2011 Oct;4(5):622-9. doi: 10.1161/CIRCEP.111.962928. Epub 2011 Aug 15. PMID 21844156